CLINICAL TRIAL: NCT04821102
Title: Investigator Initiated Trial to Evaluate Cartilage Regeneration by Arthroscopy in Patients With K-L Grade III Knee Osteoarthritis After JOINTSTEM Administration
Brief Title: Investigator Initiated Trial to Evaluate Cartilage Regeneration by Arthroscopy After JOINTSTEM Administration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: R-Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BS-JS-IIT1
Record Dates: First submitted 2021-03-24; First posted 2021-03-29 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Degenerative Arthritis; Knee Arthritis
Keywords: Stem cell; Adipose tissue derived mesenchymal stem cell; Osteoarthritis; degenerative arthritis; Biostar; Rbio
MeSH Terms: conditions — Osteoarthritis | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JOINTSTEM (Experimental): Autologous Adipose Tissue derived MSCs
  Interventions: Biological: JOINTSTEM
- Saline (Placebo Comparator): saline
  Interventions: Drug: Saline

INTERVENTIONS:
Biological: JOINTSTEM — JOINTSTEM Autologous Adipose Tissue derived MSCs 1x10^8cells/(saline), 1 time injection under ultrasonic guided
  Other Names: Autologous Adipose Tissue derived MSCs
  Arms: JOINTSTEM
Drug: Saline — saline, 1 time injection under ultrasonic guided
  Arms: Saline

SUMMARY:
The purpose of this study is to confirm cartilage regeneration through arthroscopy after a single administration of autologous Adipose Tissue derived Mesenchymal stem cells(JOINTSTEM) in patients with degenerative arthritis of K-L grade 3

DETAILED DESCRIPTION:
JOINTSTEM is injectables for an OA treatment that uses autologous adipose-derived mesenchymal stem cells. As it does not use allogenic tissues and is cultured without additional genetic modification, it is classified as 'autologous cell therapy' and is completely free of immunologic rejection.

It primarily aims to regenerate cartilage. The intra-articular injection of JOINTSTEM is expected to stimulate the regeneration of cartilage, and to innovatively improve joint function with cartilage regeneration.

The subjects of this therapy were patients with K&L grade 3 aged 20 or older.

This study is a double-blind, randomized, placebo controlled study with two arms to evaluate JOINTSTEM as a treatment for subjects with osteoarthritis. Following a 2-week screening period, approximately 21 patients will be randomly assigned into one of the following two arms in a 2:1 ratio (2 JointStem : 1 placebo control). After each patient completes 12-month visit (Visit 6) and the data management team confirms all data have no issue, the individual database will be locked and the blinding will be open for the statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20 and older, male and female
2. Patients must consent in writing to participate in the study by signing and dating an informed consent document
3. Diagnosis of degenerative arthritis of class 1-3 by ACR(American College of Rheumatology Criteria) Global functional criteria
4. Diagnosis of Kellgren and Lawrence grade 3 by radiographic criteria
5. Patients suitable for one of three conditions of 'diagnostic criteria for osteoarthritis of knee' based on ACR guideline

   * clinical and inspectional opinion
   * clinical and radiographic opinion
   * clinical opinion
6. Patients who has joint pain ≥ 50mm on 100mm VAS (Visual Analog Scale) at Screening
7. Patient who has WOMAC score ≥ 1000 at Screening
8. No improvement with persisting knee pain at least for 12 weeks (3 months) by nonoperational therapy before Screening

Exclusion Criteria:

1. Patients who have pregnancy plans within this trial period or childbearing age patients who do not agree to maintain contraception status through appropriate contraception methods

   * Appropriate contraception method: Use of condom, contraceptive sponges, foam, diaphragm, intrauterine device etc.
   * Periodic abstinence(e.g. methods of predicting ovulation) and moderation are not considered as appropriate contraception method.
   * Not allowed to use hormonal contraceptives
   * Childbearing age female patients, exclude menopausal female (amenorrhea for more than 24 months after the last menstruation) or female who has no possibility of pregnency by surgical sterilization operation, can participate in this study only determined negative in pregnancy test
2. Pregnant women or lactating mothers
3. Patients with Body Mass Index (BMI) > 35
4. Patients with positive human immunodeficiency (HIV), hepatitis B (HBV), hepatitis C (HCV), syphilis at screening indicative of current of pass infection
5. Patients with other disease including

   * Septic arthritis, Rheumatoid or Inflammatory joint disease, Gout, Reccurent pseudogout, Paget disease, Articular fractures, Ochronosis, Acromegaly, Hemochromatosis, Wilson's disease,Osteochondromatosis, Hereditary disorder, Genetic disorder of collagen
6. Patients who are diagnosed with malignant tumor in the past or present
7. Patients who have clinically significant diseases including

   * Cardiac disorder (Myocardial infarction, Coronary artery bypass graft, Arrhythmia and other severe Cardiac disorder etc.)
   * Resistant hypertension (systolic blood pressure > 160mmHg or diastolic pressure > 100mmHg at Screening)
   * Kidney disease (Chronic renal failure, Glomerulonephritis etc.)
   * Liver disease (Hepatocirrhosis, Fatty liver, acute or chronic liver disease etc.)
   * Endocrinopathy (Thyroiditis, Diabetes insipidus, Cushing disease etc.)
8. Patients who have significant lab abnormalities
9. Patients who have severe pain in other areas that can affect the judgement of knee joint symptom
10. Patients who underwent any arthroscopic surgery on the injection site within 6 months of the screening visit date, or scheduled to perform any surgery during the clinical trial period
11. Patients who received any drug by intra-articular injection(hyaluronic acid or steroid etc.) for treatment within 6 months prior to Screening
12. Patients who experienced as stem cell therapy or blood product injection(PRP, Prolo therapy etc.)
13. Patients who received treatment within 14 days prior to Screening including(But, patients who had wash-out-period can participate in this study)

    * Take medicines including composition of Glucosamine, Chondretin sulphate and Diacerhein etc.
    * Take phytotherapeutic agent or Chinese medicine for osteoarthritis
    * Take antiinflammatory analgesic drug, NSAIDs (prescription/nonprescription pharmaceuticals) etc. (Patients who have 3 days of wash-out-period after they took acetaminophen can participate in the study)
    * Take oral steroids
14. Patients with penicillin hypersensitivity reactions
15. Patients with skin diseases or infections in the area of the injection site
16. Patients who have abnormal flail over grade 2 flail knee test of anterior to posterior and varus/valgus lesion at physical examination
17. Patients who have difficulty in taking MRI because of metal materials (cardiac pacemaker or clip of cerebral artery etc.) in their body or claustrophobia -but, patients with metal materials that are not affected by magnetic field can participate in this study
18. Patients who have difficulty in liposuction or local anesthesia
19. Patients who have alcohol, drug abuse history
20. Patients who have severe neurologic and psychiatric disorders that affect clinical trials
21. Patients who had participated in other clinical trials within 12 weeks prior to this study
22. Patients who the principal investigator considers inappropriate for the clinical trial due to any other reasons than those listed above

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Arthroscopy | 48 Weeks
  Change of damaged cartilage defects after 48 weeks from IP administration, compared to Baseline (Experimental group vs Control group)

SECONDARY OUTCOMES:
WOMAC total score | 12 weeks, 24 weeks, 48 weeks
  Change of Western Ontario and McMaster Universities Osteoarthritis Index(WOMAC) total scores from baseline (Experimental group vs Control group)
WOMAC subscale score | 12 weeks, 24 weeks, 48 weeks
  Change of Western Ontario and McMaster Universities (WOMAC) subscale score (3 sub-scales: Pain, stiffness, and physical function of the knee) from baseline (Experimental group vs Control group)
VAS score | 12 weeks, 24 weeks, 48 weeks
  Change of Visual Analog Scale (VAS) from baseline (Experimental group vs Control group) Pain of knee will be measured by the 100mm VAS Score range is from 0mm(no pain) to 100mm(severe pain) Pain of knee will be measured by the 100mm Visual Analog Scale (VAS)
RAND-36 | 12 weeks, 24 weeks, 48 weeks
  Change of The RAND-36 Measure of Health-Related Quality of Life (RAND-36) score from baseline (Experimental group vs Control group) Scoring the RAND 36-Item Health Survey is a two-step process. First, precoded numeric values are recoded per the scoring key given in Table 1. Note that all items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved. In step 2, items in the same scale are averaged together to create the 8 scale scores.
IKDC | 12 weeks, 24 weeks, 48 weeks
  Change of International Knee Documentation Committee (IKDC) score from baseline (Experimental group vs Control group) The IKDC is a patient-completed tool, which contains sections on knee symptoms (7 items), function (2 items), and sports activities (2 items). Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).
Biopsy | 48 Weeks
  Change of Biopsy from baseline (Experimental group vs Control group)
Use of rescue medication | 4 Weeks, 12 Weeks, 24 Weeks, 48 Weeks
  Frequency and total amount of rescue medication administration will be measured.
Kellgren-Lawrence grade | 24 Weeks, 48 Weeks
  Change from baseline in Kellgren-Lawrence grade of knee osteoarthritis determined by X-ray at Week 48

CONTACTS AND LOCATIONS:
Overall Officials: CHANGMIN LEE, M.D.,Ph.D., Principal Investigator — Bethesda Hospital
Locations (1):
- Bethesda Hospital, Yangsan, South Korea

IPD SHARING:
Plan to Share IPD: No